CLINICAL TRIAL: NCT05548894
Title: Comparison Between the Efficacy of Stabilization Splint and Low Level Laser Therapy for Treatment of Patients With Chronic Closed Lock of the Non-reducible Temporo-mandibular Joint Disc. A Parallel Randomized Clinical Trial.
Brief Title: Comparison Between Splint and Laser in Patients Without Disc Displacement With Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: A34080622
Record Dates: First submitted 2022-09-11; First posted 2022-09-22 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-08

CONDITIONS: TMJ Disc Disorder
MeSH Terms: interventions — Laser Therapy; Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Parallel clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- stabilization splint (Active Comparator): acrylic splint in the maxillary arch with flat surface
  Interventions: Device: stabilization splint
- laser therapy (Active Comparator): laser beam directed to the affected part cause activation of blood circulation
  Interventions: Device: laser therapy
- stabilization splint and laser therapy (Active Comparator): using both laser therapy and stabilization splint for more improvement
  Interventions: Device: stabilization splint and laser therapy

INTERVENTIONS:
Device: stabilization splint — upper acrylic splint rest on the maxillary teeth and had flat surface
  Other Names: upper acrylic full arch splint
  Arms: stabilization splint
Device: laser therapy — The laser apparatus had a hand piece on which either a specially designed optic prism was attached to transfer laser energy to the tip of the prism
  Other Names: Low-level laser therapy
  Arms: laser therapy
Device: stabilization splint and laser therapy — the stabilization splint used in combination of treatment with laser therapy
  Other Names: splint combined with low level laser therapy
  Arms: stabilization splint and laser therapy

SUMMARY:
Stabilization splint therapy and Low-level laser therapy may serve as non-invasive intervention for painful temporomandibular disorders, but its efficacy is still debated. This study compared the effect of stabilization splint and low-level laser therapy alone or in combination in patients with painful chronic closed lock of temporomandibular joints disc displacement without Reduction 42 patients diagnosed with chronic closed lock of disc displacement without reduction were allocated equally and randomly into three treatment groups: group I received combined stabilization splint and low- level laser therapy, group II received low - level laser therapy and group III received stabilization splint. They were evaluated at baseline and one week, two weeks, four weeks, three months, and six months after the intervention.

DETAILED DESCRIPTION:
Objectives: Stabilization splint therapy and low- level laser therapy may serve as non-invasive intervention for painful temporomandibular disorders, but its efficacy is still debated. This study compared the effect of stabilization splint and low- level laser therapy alone or in combination in patients with painful chronic closed lock of temporomandibular joints disc displacement without Reduction.

Patients and methods: 42 patients diagnosed with chronic closed lock of disc displacement without reduction were allocated equally and randomly into three treatment groups: group I received combined stabilization splint and low-level laser therapy, group II received low-level laser therapy and group III received stabilization splint. They were evaluated at baseline and one week, two weeks, four weeks, three months, and six months after the intervention. Time of being normal was also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic closed lock patients
* Must not be able to open their mouth

Exclusion Criteria:

* neurologic diseases
* TMJ pathologic lesions

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-02-06 (Actual); Study Completion 2022-03-06 (Actual)

PRIMARY OUTCOMES:
evaluation of mouth opening | 6 months
  improvement in mouth opening or not
Masticatory muscles palpation | 6 months
  the masticatory muscles were palpated bilaterally with firm and constant pressure of one kg lasted two seconds to define painful areas
temporomandibular joint palpation | 6 months
  joint pain was achieved by first palpating the temporomandibular joint lateral pole by placing the index finger with firm and constant pressure of half kg lasted
  two seconds over the condyle in front of the tragus

CONTACTS AND LOCATIONS:
Overall Officials: Noha Elshahid, Principal Investigator — lecturer at mansoura university prosthodontic department
Locations (1):
- Mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ooi K, Yura S, Inoue N, Totsuka Y. Factors related to the incidence of anterior disc displacement without reduction and bony changes of the temporomandibular joint in patients with anterior open bite. Oral Maxillofac Surg. 2014 Dec;18(4):397-401. doi: 10.1007/s10006-013-0424-3. Epub 2013 Jul 9. PMID 23835639
- [Background] Samdal F, Amland PF, Sandsmark M, Hall C, Aasen AO. Suction-assisted lipectomy does not increase the risk of random flap necrosis in a randomized study in pigs. Aesthetic Plast Surg. 1995 Nov-Dec;19(6):549-53. doi: 10.1007/BF00454320. PMID 8638492
- [Derived] El-Shaheed NH, Mostafa AZH, Aboelez MA. Efficacy of stabilisation splint and low-level laser therapy for patients with chronic closed lock from non-reducible displaced temporo-mandibular joint discs: A parallel randomised clinical trial. J Oral Rehabil. 2023 Mar;50(3):177-193. doi: 10.1111/joor.13405. Epub 2023 Jan 5. PMID 36564950